CLINICAL TRIAL: NCT03733574
Title: A Randomized, Open-Label, 2-Treatment, 2-Sequence, 2-Period Crossover Trial to Assess the Bioequivalence of 80 mg LY03005 to 50 mg Pristiq After Single Dose Administration Under Fasting Conditions to Healthy Subjects
Brief Title: A Study of LY03005 vs Pristiq
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY03005/CT-USA-106
Record Dates: First submitted 2018-07-24; First posted 2018-11-07 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Disorder
Keywords: Depressive Disorder, Major; Depressive Disorder; Mood Disorders; Mental Disorders; Desvenlafaxine Succinate; Serotonin and Noradrenaline Reuptake Inhibitors; Neurotransmitter Uptake Inhibitors; Membrane Transport Modulators; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Physiological Effects of Drugs; Antidepressive Agents; Psychotropic Drugs
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Mood Disorders; Mental Disorders | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY03005 cross-over to Pristiq® (Desvenlafaxine) (Experimental): Subjects in this group will receive an 80 mg oral dose of LY03005. After a washout period of up to 4 days, the subjects will be switched and will receive a 50 mg oral dose of desvenlafaxine (Pristiq®).
  Interventions: Drug: LY03005; Drug: Pristiq
- Pristiq® (Desvenlafaxine) cross-over to LY03005 (Experimental): Subjects in this group will receive a 50 mg oral dose of desvenlafaxine (Pristiq®) After a washout period of up to 4 days, the subjects will be switched and will receive an 80 mg oral dose of LY03005
  Interventions: Drug: LY03005; Drug: Pristiq

INTERVENTIONS:
Drug: LY03005 — Drug: LY03005 80 mg, oral tablets, single dose
Drug: Pristiq — Drug: Pristiq 50 mg, oral tablets, single dose
  Other Names: Desvenlafaxine

SUMMARY:
The objective of this study is to evaluate relative bioavailability between 80 mg LY03005 oral tablets and 50 mg Pristiq® oral tablets after a single dose of each drug in a cross-over 2-period design under fasting condition in healthy subjects between 18 and 50 years of age.

DETAILED DESCRIPTION:
Fifty six (56) eligible subjects will be enrolled and assigned to either Group A or Group B at a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent and complying with trial procedures;
2. Male and female subjects between the ages of 18 and 50 years, inclusive;
3. Considered healthy by the Investigator based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
4. Nonsmoker, defined as not having smoked or used any form of tobacco for at least 6 months before Screening based on subject report;
5. Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight not less than 50 kg;
6. Willing and able to adhere to trial procedures and to be confined at the clinical research unit (CRU).
7. All female subjects (childbearing potential and non-childbearing potential) must have a negative serum pregnancy test result at Screening. In addition, female subjects must meet 1 of the following 3 conditions: (i) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal occlusion) based on subject report, or (iii) if of childbearing potential and heterosexually active, practicing or agree to practice a highly effective method of contraception. Highly effective methods of birth control include an intrauterine device (IUD), intrauterine hormone-releasing system (IUS), and contraceptives (oral, skin patches, or implanted or injectable products) using combined or progestogen-only hormonal contraception associated with inhibition of ovulation. A vasectomized male partner is an acceptable birth control method if the vasectomized partner is the sole sexual partner of the female subject and the vasectomized partner has received medical confirmation of surgical success.

Highly effective methods of birth control must be used for at least 14 days prior to study drug dosing, through the end of study (EOS) visit or early termination, and for a minimum of 1 month after the last dose of study drug to minimize the risk of pregnancy. Sexually active, fertile, male subjects must be willing to use acceptable contraception methods (such as double-barrier methods of a combination of male condom with either cap, diaphragm, or sponge with spermicide) from the first dose of study drug through the EOS visit or early termination, and for a minimum of 1 month after the last dose of study drug.

Exclusion Criteria:

1. Clinically significant past medical history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric (including life-long history of depression and/or anxiety), renal, hepatic, bronchopulmonary, neurologic, immunologic, ophthalmological, or lipid metabolism disorders; or drug hypersensitivity; or any other condition that in the judgement of the Investigator will affect the trial results or the subject's safety;
2. History of suicide attempt in the past 12 months and/or seen by the Investigator as having a significant history of risk of suicide or homicide;
3. History or presence of malignancy other than adequately treated and cured basal cell carcinoma or squamous cell carcinoma (skin cancer);
4. Clinically relevant illness within 1 month prior to Screening or at Screening that may interfere with the conduct of this trial;
5. Medically uncontrolled high blood pressure with mean systolic blood pressure >140 mmHg or mean diastolic blood pressure >90 mmHg at Screening after 3 measurements (after at least 5 minutes of rest in a seated position);
6. History of Long QT Syndrome (LQTS) or a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
7. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
8. History of seizure (history of febrile seizure allowed);
9. Hospital admission or major surgery within 30 days prior to Screening;
10. Participation in any other investigational drug trial within 30 days prior to Screening;
11. History of prescription drug abuse or illicit drug use within 6 months prior to Screening;
12. History of alcohol abuse according to medical history within 6 months prior to Screening;
13. Positive screen for alcohol and/or drugs of abuse;
14. Tobacco use within 6 months prior to Screening based on positive nicotine screen;
15. History of intolerance or hypersensitivity to ODV or medicines containing ODV or its precursor venlafaxine;
16. Participation in a previous clinical trial of either LY03005 or ODV or medicines containing ODV or its precursor, venlafaxine, within 30 days prior to Screening;
17. Unwillingness or inability to comply with food and beverage restrictions during trial participation;
18. Donation of blood of more than 1 unit (approximate 450 mL) or blood products or acute loss of blood during the 90 days prior to Screening;
19. Use of prescription or over-the-counter (OTC) medications and/or herbals (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at <3g/day is permitted until 24 hours prior to dosing).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
concentration-time curve (AUC) | 15 days
  Plasma ODV area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Sun, MD, PhD, MBA, Study Chair — Luye Pharma Group Ltd.
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Drug information — http://druginfo.nlm.nih.gov/drugportal/
- See also: Desvenlafaxine — http://druginfo.nlm.nih.gov/drugportal/name/Desvenlafaxine
- See also: Desvenlafaxine Succinate — http://druginfo.nlm.nih.gov/drugportal/name/desvenlafaxine%20succinate
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks
- See also: Pristiq (Desvenlafaxine) Label - FDA — http://www.accessdata.fda.gov/drugsatfda_docs/label/2012/021992s030lbl.pdf